CLINICAL TRIAL: NCT02141451
Title: Study of the ADAM17 Inhibitor INCB7839 Combined With Rituximab After Autologous Hematopoietic Cell Transplantation (HCT) For Patients With Diffuse Large B Cell Non-Hodgkin Lymphoma (DLBCL)
Brief Title: ADAM17 Inhibitor/ Rituximab After Auto HCT for DLBCL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2013LS081; HM2013-24 (Other: University of Minnesota Blood and Marrow Transplant Program)
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Results first posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Diffuse Large B Cell Non-Hodgkin Lymphoma
Keywords: DLBCL
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: A Fast-Track Design with 1 patient enrolled per dose level until a grade 2 or greater treatment emergent adverse event occurs. A treatment emergent adverse event is any event not present prior to the initiation of the treatment (INCB7839) or any event already present that worsens in either intensity or frequency following exposure to the treatment. At that point, dose escalation will convert to a standard 3+3 design with two additional patients enrolled at the same dose level. If dose level 3 is completed without dose limiting toxicity (DLT) in the 1st 3 patients, an additional 3 patients will be enrolled at this level (without the staggering required by the DLT rules) prior to moving to the phase II component.
  Once the phase I dose escalation is completed, an additional 12 patients will be enrolled at the MTD (or dose level 300mg bid, if no DLT) to obtain a more detailed toxicity profile as well as a preliminary estimate of progression free survival at 6 months post-transplant.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- INCB7839 100 mg (Phase I) (Experimental): Rituximab will be given after day +28 re-staging and again 1 and 7 weeks later, followed by INCB7839 at assigned dose twice daily for 90 days - begin the morning of the 2nd dose of rituximab Rituximab: Rituximab 375 mg/m2 IV after day +28 (as late as day 75) re-staging and again 1 and 7 weeks later INCB7839: INCB7839 at assigned dose twice daily for 90 days - begin the morning of the 2nd dose of rituximab
  Interventions: Drug: Rituximab; Drug: INCB7839
- INCB7839 200 mg (Phase I) (Experimental): Rituximab will be given after day +28 re-staging and again 1 and 7 weeks later, followed by INCB7839 at assigned dose twice daily for 90 days - begin the morning of the 2nd dose of rituximab Rituximab: Rituximab 375 mg/m2 IV after day +28 (as late as day 75) re-staging and again 1 and 7 weeks later INCB7839: INCB7839 at assigned dose twice daily for 90 days - begin the morning of the 2nd dose of rituximab
  Interventions: Drug: Rituximab; Drug: INCB7839
- INCB7839 300 mg (Phase I) (Experimental): Rituximab will be given after day +28 re-staging and again 1 and 7 weeks later, followed by INCB7839 at assigned dose twice daily for 90 days - begin the morning of the 2nd dose of rituximab Rituximab: Rituximab 375 mg/m2 IV after day +28 (as late as day 75) re-staging and again 1 and 7 weeks later INCB7839: INCB7839 at assigned dose twice daily for 90 days - begin the morning of the 2nd dose of rituximab
  Interventions: Drug: Rituximab; Drug: INCB7839
- INCB7839 (Phase II) (Experimental): Rituximab will be given after day +28 re-staging and again 1 and 7 weeks later, followed by INCB7839 at assigned dose twice daily for 90 days - begin the morning of the 2nd dose of rituximab Rituximab: Rituximab 375 mg/m2 IV after day +28 (as late as day 75) re-staging and again 1 and 7 weeks later INCB7839: INCB7839 at assigned dose twice daily for 90 days - begin the morning of the 2nd dose of rituximab
  Interventions: Drug: Rituximab; Drug: INCB7839

INTERVENTIONS:
Drug: Rituximab — Rituximab 375 mg/m2 IV after day +28 (as late as day 75) re-staging and again 1 and 7 weeks later
  Other Names: Rituxan
Drug: INCB7839 — INCB7839 at assigned dose twice daily for 90 days - begin the morning of the 2nd dose of rituximab

SUMMARY:
This is a single institution phase I/II study using an ADAM17 inhibitor (INCB7839) with rituximab as consolidation therapy after an autologous hematopoietic cell transplant (HCT) for patients with diffuse large B cell lymphoma (DLBCL). The study consists of two phases. The dose finding phase is a modified version of a phase I trial and the extended phase is a modified version of a phase II trial.

DETAILED DESCRIPTION:
The primary goal of the dose finding phase is to determine the maximum tolerated dose (MTD) of INCB7839. Up to three dose levels will be tested (100 mg bid, 200 mg bid, and 300 mg bid). As the 300 mg bid has been proven safe in the non-transplant setting, dose escalation follows a Fast-Track Design with 1 patient enrolled per dose level unless a grade 2 or greater treatment emergent event occurs within the 1st 14 days of INCB7839. At that point, dose escalation converts to a standard 3+3 design and two additional patients are enrolled at the current dose level. If dose level 3 is completed without dose limiting toxicity (DLT) in the 1st 3 patients, an additional 3 patients will be enrolled at this level (without the staggering required by the DLT rules) prior to moving to the phase II component.

Once the phase I dose escalation is completed, an additional 12 patients will be enrolled at the MTD (or dose level 3, if no DLT) to obtain a more detailed toxicity profile as well as a preliminary estimate of progression free survival at 6 months post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older who have undergone an autologous HCT for the treatment of DLBCL and are in a complete remission (CR), partial remission (PR) or have stable disease (SD) at the day 28 post-transplant reassessment
* Karnofsky Score of ≥ 70% (appendix II)
* Able to start the protocol therapy (1st dose of rituximab) between day 28-75 post-transplant
* Adequate organ function defined as:

  * Hematologic: platelets ≥ 50,000 x 109/L; ANC ≥ 1000 x 109/L unsupported by G-CSF or GM-CSF for 3 days
  * Renal: creatinine < 1.5 mg/dl or glomerular filtration rate > 50 ml/min
  * Hepatic: Alanine transaminase (ALT, SGPT) and aspartate aminotransferase (SGOT, AST) < 3 x upper limit of institutional normal and total bilirubin < 3.0 mg/dl (if total bilirubin is ≥ 3.0 patient is eligible if direct bilirubin is within normal limits)
  * Pulmonary: clinically no evidence of pulmonary disease
  * Cardiac: no symptoms of uncontrolled cardiac disease
* If post-transplant consolidation radiation therapy is given, the patient must be at least 14 days between last radiation treatment and 1st dose of rituximab
* Able to take daily aspirin (325 mg) for the duration of INCB7839 treatment and 1 week after the last dose to reduce the risk of thrombosis (not applicable if on other anti-coagulant therapy at time of study enrollment)
* Females are either postmenopausal for at least 1 year, are surgically sterile for at least 3 months, or must agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through 12 months after the last dose of rituximab if of childbearing potential. (Note: Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the participants and their understanding confirmed).
* Males must agree to take appropriate precautions to avoid fathering a child (with at least 99% certainty) from screening through 12 months after the last dose of rituximab. (Note: Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the participants and their understanding confirmed).
* Voluntary written consent signed before performance of any study-related procedure not part of normal medical care

Exclusion Criteria:

* Pregnant or lactating - Studies to evaluate the potential for embryo toxicity and teratogenicity have not been performed for INCB7839. Until additional information is available, women of childbearing potential should use appropriate precautions to avoid becoming pregnant. Rituximab is Pregnancy Category C: There are no adequate and well-controlled studies of rituximab in pregnant women. Females of childbearing potential must have a negative urine or serum pregnancy test within 14 days of study treatment start
* Recent venous thrombosis within 4 weeks prior to study enrollment. Patients at high risk for thrombotic events due to inherited risk factors (i.e. factor V Leiden) or DVT/PE in the past 12 months should be on secondary prophylaxis with anti-coagulant therapy (i.e. warfarin or low molecular weight heparin) prior to enrollment
* Active uncontrolled infection
* Active CNS disease
* Previous severe or life-threatening allergic reaction with rituximab or known allergy to the compounds found in INCB7839
* Any gastrointestinal condition causing malabsorption or obstruction (eg, celiac sprue, gastric bypass surgery, strictures, adhesions, history of small bowel resection, blind loop syndrome)
* Unwilling or unable to swallow tablets BID
* Serologic or clinical evidence of current active hepatitis B or C infection, defined as elevated levels of Hep B antigen or Hep C antibody (unless active infection is ruled out by nucleic acid tests)
* Known HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2019-01-23 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Bachanova, MD, Principal Investigator — University of Minnesota Medical Center, Fairview
Locations (1):
- University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- INCB7839 300 mg (Phase II): Rituximab will be given after day +28 re-staging and again 1 and 7 weeks later, followed by INCB7839 at assigned dose twice daily for 90 days - begin the morning of the 2nd dose of rituximab
  Rituximab: Rituximab 375 mg/m2 IV after day +28 (as late as day 75) re-staging and again 1 and 7 weeks later
  INCB7839: INCB7839 at assigned dose twice daily for 90 days - begin the morning of the 2nd dose of rituximab
Period: Overall Study
Arm/Group | INCB7839 100 mg (Phase I) | INCB7839 200 mg (Phase I) | INCB7839 300 mg (Phase I) | INCB7839 300 mg (Phase II)
Started | 3 | 4 | 7 | 16
Completed | 3 | 2 | 2 | 7
Not Completed | 0 | 2 | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | INCB7839 100 mg (Phase I) | INCB7839 200 mg (Phase I) | INCB7839 300 mg (Phase I) | INCB7839 300 mg (Phase II) | Total
Number analyzed (Participants) | 3 | 4 | 7 | 16 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 4 | 10 | 20
  >=65 years | 0 | 1 | 3 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.67 (4.78) | 59.25 (8.79) | 53.86 (14.67) | 57.19 (11) | 56.93 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 7 | 13
  Male | 0 | 3 | 5 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 7 | 16 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 4 | 7 | 16 | 30
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity Events
Description: The Phase I design will continue until the MTD is declared or until the first dose is declared to be above MTD. Phase I dose limiting toxicity (DLT) is defined as Grade 3-5 non-hematologic, non-infectious toxicity including thromboembolic complications and select hematologic events including: grade 4 neutropenia lasting for ≥ 7 days, febrile neutropenia, grade 4 thrombocytopenia lasting ≥ 7 days despite dose delay or grade 3 thrombocytopenia associated with bleeding.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | INCB7839 100 mg (Phase I) | INCB7839 200 mg (Phase I) | INCB7839 300 mg (Phase I)
Number analyzed (Participants) | 3 | 4 | 7
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Progression Free Survival at 6 Months
Description: This primary end point will be estimated with Kaplan-Meier curves.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | INCB7839 100 mg (Phase I) | INCB7839 200 mg (Phase I) | INCB7839 300 mg (Phase I) | INCB7839 300 mg (Phase II)
Number analyzed (Participants) | 3 | 4 | 7 | 16
Participants | 3 | 3 | 6 | 15

3. Secondary Outcome: Incidence of Serious Adverse Events
Description: To determine incidence of serious adverse events
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | INCB7839 100 mg (Phase I) | INCB7839 200 mg (Phase I) | INCB7839 300 mg (Phase I) | INCB7839 300 mg (Phase II)
Number analyzed (Participants) | 3 | 4 | 7 | 16
Participants | 0 | 0 | 1 | 3

4. Secondary Outcome: Overall Survival
Description: To evaluate 1 year overall survival
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | INCB7839 100 mg (Phase I) | INCB7839 200 mg (Phase I) | INCB7839 300 mg (Phase I) | INCB7839 300 mg (Phase II)
Number analyzed (Participants) | 3 | 4 | 7 | 16
Participants | 3 | 3 | 7 | 16

5. Secondary Outcome: Time to Progression
Description: Time to relapse/progression in days
Time Frame: 1 year
Population: Only 3 participants experienced disease progression by 1 year on study
Measure: Number; unit: days
Arm/Group | INCB7839 100 mg (Phase I) | INCB7839 200 mg (Phase I) | INCB7839 300 mg (Phase I) | INCB7839 300 mg (Phase II)
Number analyzed (Participants) | 0 | 1 | 1 | 1
days |  | 105 | 136 | 259

ADVERSE EVENTS:
Time Frame: 105 days or 1 week after last dose of INCB7839 if it is discontinued earlier
Arm/Group | INCB7839 100 mg (Phase I) | INCB7839 200 mg (Phase I) | INCB7839 300 mg (Phase I) | INCB7839 300 mg (Phase II)
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/4 | 2/7 | 2/16
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 1/7 | 3/16
Other Adverse Events (participants affected / at risk) | 3/3 | 3/4 | 7/7 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INCB7839 100 mg (Phase I) (N=3) | INCB7839 200 mg (Phase I) (N=4) | INCB7839 300 mg (Phase I) (N=7) | INCB7839 300 mg (Phase II) (N=16)
Norovirus and C-Diff (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INCB7839 100 mg (Phase I) (N=3) | INCB7839 200 mg (Phase I) (N=4) | INCB7839 300 mg (Phase I) (N=7) | INCB7839 300 mg (Phase II) (N=16)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Alkaline phosphate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic Reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (4) | 7 (9)
Arthalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
D-dimer increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (15)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leg cramps (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restless legs / leg pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (hands) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C. difficile (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shingles (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection - HSV (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection - VZV (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
D-dimer increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (15) | 2 (3) | 1 (5) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 8 (12)
Neutrophil count decreased (Investigations) | 3 (5) | 1 (2) | 1 (2) | 4 (6)
Pain (General disorders) | 0 (0) | 1 (1) | 2 (2) | 6 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 3 (4) | 3 (10)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash-pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vital capacity abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (5)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
White blood cell decreased (Investigations) | 3 (8) | 1 (2) | 1 (1) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/51/NCT02141451/Prot_SAP_000.pdf